CLINICAL TRIAL: NCT06938087
Title: Pilot Study to Assess Safety and Performances of a Energy Storing and Return (ESAR) Prosthetic Foot Made in Additive Manufacturing
Brief Title: Assessment of Safety and Performances of a 3D Printed Prosthetic Foot: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Collaborators: Istituto per i Polimeri Compositi e Biomateriali (CNR-IPCB) (Unknown); Istituto di Chimica della Materia Condensata e di Tecnologie per l'Energia (CNR-ICMATE) (Unknown)
Responsible Party: Principal Investigator, Emanuele Gruppioni, Engineer, Orthopaedic Techinician, Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-PAI-01-23
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Amputation of Lower Limb
Keywords: Safety; Lower limb amputation; Additive manufacturing; Prosthesis foot; Performances

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROFIL prosthesis foot (Experimental): Recruited subjects with below kenen amputation wearing the experimental prosthesis foot (PROFIL)
  Interventions: Device: 3D printed prosthesis foot
- Current prosthesis foot (PROFLEX XC) (Active Comparator): Recruited subjects with below knee amputation wearing the currently used prosthesis foot (PROFIL)
  Interventions: Device: Current prosthesis foot

INTERVENTIONS:
Device: 3D printed prosthesis foot — Energy storage and restoration 3D printed prosthesis foot
  Arms: PROFIL prosthesis foot
Device: Current prosthesis foot — Energy storage and restitution prosthesis foot made in carbon fibers blades
  Arms: Current prosthesis foot (PROFLEX XC)

SUMMARY:
A dynamic energy storage and return foot prosthesis is a type of prosthesis designed to mimic and restore the functionality and natural movement of the limb that has been amputated. This type of prosthesis is designed to allow patients to perform daily activities, even very dynamic ones, with greater ease and efficiency. The distinguishing feature of a dynamic energy storage and return prosthesis is the presence of a system that accumulates mechanical energy during the support phase on the ground and returns it during the push phase, increasing the amount of push itself. In foot prostheses, it is common to use carbon fiber blades or springs that deform during the support of the foot and then restore themselves, returning elastic energy during the subsequent push. This helps reduce the effort required to walk and allows for more fluid and natural movements. Additive Manufacturing (AM) technology is ideal for highly customized and high-value production. Orthoses/prostheses are particularly suited to exploit the potential of this technology. However, the lack of functional materials that meet different design needs, such as structure and comfort of the devices, has limited the use of AM mainly in orthoses. AM is promising for orthoses due to its customization capability and reduced production costs compared to traditional solutions. In particular, it has been shown how continuous filament carbon printing can lead to the creation of prostheses that have dynamic and energy return characteristics similar to or even superior to commercial ones. The present pilot clinical investigation aims to provide indications regarding the safety and performance of the 3D printed prosthesis - named PROFIL - in a real-world scenario. The state of the art has not yet defined the performance and safety of 3D printed prostheses with thermoplastic materials and continuous carbon fiber. Since greater comfort and the possibility of performing physical activity more easily with the use of these devices is expected, it is considered of interest for clinical practice to evaluate these prostheses. The primary objective of the study is therefore to evaluate the safety and performance of the device during walking on flat surfaces and more demanding tasks. The secondary objectives aims at evaluate usability and deformation of the 3D printed prosthesis under different loading conditions (slow and fast walking, ascending and descending ramps or steps) by mean of fiber-glass sensors integrated in the prosthesis foot.

ELIGIBILITY:
Inclusion Criteria:

* Monolateral below knee amputation
* Mobility level: K3 or K4
* Age: 18-65 years old
* Maximum weigth: 100 Kg
* Collaborative subject
* Clinically stable stump

Exclusion Criteria:

* Pregnant
* Not able to understand written and oral instructions
* Problems to the stump

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-04-17 (Estimated); Study Completion 2025-04-17 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events occurred during use of the Intervention prosthesis foot | Day 1 and Day 2
  Adverse events may be: falling, stumbling, lower back pain as consequence of the prosthesis foot use, stump pain as consequence of the prosthesis foot use, breakage of the prosthesis foot
Change from Comparator of joints kinematics measured with Inertial Measurements Units (IMUs) placed on subject lower leg, upper arms and trunk | Day 1 and Day 2
  The IMUs record subject's joints kinematics while performing a series of motor tasks, i.e. walk of flat surfaces at a self-selected speed and ascend/descend stairs and ramps.
Change from Comparator of joints kinematics and dymamics measured with an optoelectronic system | Day 1 and Day 2
  The optoelectronic system records subject's joints kinematics and dynamics during subject's walk on a flat surface at a self-selected speed.
Change from Comparator of gait quality wihile ascending ramps with Hill Assessment Index (HAI) | Day 1 and Day 2
  HAI is a 11-points ordinal scale; the higher the score the better the gait quality while ascending ramps
Change from Comparator of gait quality while ascending stairs with Stair Ascending Index (SAI) | Day 1 and Day 2
  SAI is 13-points ordinal scale; the higher the score the better the gait quality while ascending ramps
Change from Comparator of equilibrium in orthostatism by mean of force plates | Day 1 and Day 2
  The subject is asked to stand still on a force plate for 30 seconds. The sway of the Centre of Pressure (COP) is recorded. The higher the sway, the lower the equilibrium in orthostatism
Change from Comparator of load simmetry while standing up/sitting down from/on a chiar by mean of force plates | Day 1 and Day 2
  The subject is asked to sit on a chair with both the feets (sound foot and prosthesis foot) on different force plates. At the "Start" signal, the subject stands up, stands still for 5 seconds and sits down. The weigth distribution on the lower limbs is recorded during the entire task.
Change from Comparator of subject mobility with prosthesis by mean of the Amputee Mobility Predictor (AMP) | Day 1 and Day 2
  AMP is a 21-item objectve measure in which static and dynamic sitting and standing activities, as well as transfer and gait skills of progressing difficulty are performed. Score range is 0-47. Higher scores indicate better mobility.
Change form Comparator of functional mobility measured with the L-test | Day 1 and Day 2
  The subject starts from a sitting position. At the "Start" signal, the subject stands up from the chair, walks in a closed 10-meters L-shaped path, and sits down on the same chair. The time necessary to complete the path is measured. The lower the time, the higher the functional mobility.

SECONDARY OUTCOMES:
Change from Comparator of usability of the prosthesis foot | Day 1 and Day 2
  Usability is measured with an ad hoc custom-made questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Protesi Inail, Vigorso Di Budrio, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anthropometric characteristics Kinematics data measured via IMUs, optoelectronic system and force plates Scores of PROMs
Supporting Information: Study Protocol
Time Frame: IPD will be availabale within 6 months after study completion. Study completion is expected to occur by April 17th 2025
Access Criteria: IPD will be shared with Istituto per i Polimeri Compositi e Biomateriali (CNR-IPCB) and Istituto di Chimica della Materia Condensata e di Tecnologie per l'Energia (CNR-ICMATE), both located in Lecco (Italy). Both the Institutions contributed to the development and manufacturing of the 3D printed prosthesis foot under evaluation.

REFERENCES:
- [Background] Manero A, Smith P, Sparkman J, Dombrowski M, Courbin D, Kester A, Womack I, Chi A. Implementation of 3D Printing Technology in the Field of Prosthetics: Past, Present, and Future. Int J Environ Res Public Health. 2019 May 10;16(9):1641. doi: 10.3390/ijerph16091641. PMID 31083479
- [Background] South BJ, Fey NP, Bosker G, Neptune RR. Manufacture of energy storage and return prosthetic feet using selective laser sintering. J Biomech Eng. 2010 Jan;132(1):015001. doi: 10.1115/1.4000166. PMID 20524754
- [Background] Klute GK, Berge JS, Orendurff MS, Williams RM, Czerniecki JM. Prosthetic intervention effects on activity of lower-extremity amputees. Arch Phys Med Rehabil. 2006 May;87(5):717-22. doi: 10.1016/j.apmr.2006.02.007. PMID 16635636
- [Background] Versluys R, Beyl P, Van Damme M, Desomer A, Van Ham R, Lefeber D. Prosthetic feet: state-of-the-art review and the importance of mimicking human ankle-foot biomechanics. Disabil Rehabil Assist Technol. 2009 Mar;4(2):65-75. doi: 10.1080/17483100802715092. PMID 19253096
- [Background] Hafner BJ, Sanders JE, Czerniecki J, Fergason J. Energy storage and return prostheses: does patient perception correlate with biomechanical analysis? Clin Biomech (Bristol). 2002 Jun;17(5):325-44. doi: 10.1016/s0268-0033(02)00020-7. PMID 12084537